CLINICAL TRIAL: NCT05599061
Title: Treatment of Functionally Non-significant Vulnerable Plaques in Patients With Multivessel ST-elevation Myocardial Infarction The VULNERABLE Randomized Trial
Brief Title: Treatment of Functionally Non-significant Vulnerable Plaques in Patients With Multivessel ST-elevation Myocardial Infarction The VULNERABLE Trial
Acronym: VULNERABLE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación EPIC (Other)
Collaborators: Abbott (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: EPIC28-VULNERABLE
Record Dates: First submitted 2022-10-25; First posted 2022-10-31 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Coronary Artery Disease; Coronary Disease; Ischemic Heart Disease
Keywords: Vulnerable Plaque; Optical Coherence Tomography; Fractional Flow Reserve and ST-elevation Myocardial Infarction
MeSH Terms: conditions — Coronary Artery Disease; Coronary Disease; Myocardial Ischemia; ST Elevation Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Optimal Medical Treatment (OMT) + PCI (Experimental)
  Interventions: Other: FFR>0.80+ OCT with findings indicative of vulnerable plaque
- Optimal Medical Treatment (OMT) (Active Comparator)
  Interventions: Other: FFR>0.80+ OCT with findings indicative of vulnerable plaque

INTERVENTIONS:
Other: FFR>0.80+ OCT with findings indicative of vulnerable plaque — Patients received OPTIMAL MEDICAL TREATMENT (OMT)+PCI
  Arms: Optimal Medical Treatment (OMT) + PCI
Other: FFR>0.80+ OCT with findings indicative of vulnerable plaque — OPTIMAL MEDICAL TREATMENT (OMT)
  Arms: Optimal Medical Treatment (OMT)

SUMMARY:
The study aims to compare a preventive percutaneous coronary intervention (PCI) plus optimal medical treatment (OMT) strategy vs. OMT for treatment of non-functionally significant non-culprit lesions presenting with optical coherence tomography (OCT) findings indicative of vulnerable plaque, in patients with ST-elevation myocardial infarction (STEMI) and multivessel disease.

DETAILED DESCRIPTION:
STEMI patients with multivessel disease planned for invasive evaluation of intermediate lesions (40-69% stenosis) are initially investigated with fractional flow reserve (FFR). Patients with FFR ≤ 0.80 are considered as screening failure and treated with PCI. Patients with FFR > 0.80 are then investigated with optical coherence tomography (OCT). Patients without OCT findings of vulnerable plaque are treated with OMT and included in the OMT registry arm. Patients presenting with OCT characteristics of vulnerable plaque are included in the randomized trial comparing PCI with stent implantation plus OMT versus OMT.

ELIGIBILITY:
Inclusion Criteria:

* Patients > 18 years.
* Successful revascularization of the culprit lesion in patients undergoing coronary angiography due to ST-segment elevation (> 1mm in > 2 contiguous leads, new left bundle branch block, or true posterior MI with ST depression of >1mm in >2 contiguous anterior leads) in the first 72 hours of the symptom's onset.
* Multivessel coronary disease with non-culprit lesions located in different vessels than the culprit lesion and ranging from 40 to 69% of DS (visual estimated diameter stenosis ) by visual estimate planned for FFR-guided revascularization in staged procedure (>24 hours and <60 days after PCI of the culprit lesion).
* Non-culprit lesions should be suitable for functional assessment with pressure wire and OCT catheter and should be suitable to be treated with a single 2.0 to 4.5 mm EES (everolimus-eluting stent ).
* Subject agrees to not participate in any other clinical trial study for a period of 4 years following the inclusion in the study.
* Informed consent signed.

Exclusion Criteria:

* Inability to provide informed consent.
* Female of childbearing potential (age <50 years and last menstruation within the last 12 months), who did not undergo tubal ligation, ovariectomy or hysterectomy.
* Known intolerance to aspirin, heparin, everolimus, contrast material.
* Unresolved mechanical complication or cardiogenic shock at the staged procedure.
* Non-culprit study lesions located in the left main coronary artery or in coronary vessels with prior coronary revascularization (PCI or by-pass) or with distal vessel occlusion.
* Patients with long, bifurcated, severely angulated or severely calcified non-culprit study lesions non suitable to be treated with a single EES implantation.
* Asthma or known history of bronchial hyper-reactivity.
* Chronic renal dysfunction with creatinine clearance < 45 ml/min.
* Severe comorbidities that in the opinion of the local investigators determine the patient's life expectancy < 4 years.
* Subject is currently participating in another clinical trial that has not yet completed its primary endpoint.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2023-01-30 (Actual); Primary Completion 2028-12-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Target Vessel Failure (TVF) | 4 Years
  TVF as a composite of :
  Cardiovascular Death Target-vessel related MI Clinically and physiologically-oriented Target vessel revascularization

SECONDARY OUTCOMES:
Cardiac death | 4 Years
  To compare Cardiac death between both groups in the randomized arm death.
All-cause Death | 4 Years
  To compare all death between both groups in the randomized arm death.
All Myocardial Infarctions | 4 Years
  To compare Myocardial Infarctions between both groups in the randomized arm death. death
Target-Vessel Myocardial Infarction | 4 Years
  To compare target-vessel myocardial infarction between both groups in the randomized arm.
Revascularizations | 4 Years
  To compare all revascularizations between both groups in the randomized arm.
Ischemic-driven target vessel revascularization | 4 Years
  To compare ischemic-driven target vessel revascularization between both groups in the randomized arm.
Patient-oriented endpoint of major adverse cardiac events | 4 Years
  To compare the patient-oriented endpoint of major adverse cardiac events, a composite of all-cause death, myocardial infarction, and revascularization between both groups in the randomized arm.
Target Vessel Failure (TVF) | 4 Years
  To compare the TVF rate between patients included in the OMT group of the randomized arm (presenting with vulnerable plaque) vs. patients included in the OMT registry (without vulnerable plaque).
Fractional Flow Reserve (FFR) | 4 years
  To compare the FFR values between patients with vulnerable plaques (randomized arm) and patients without vulnerable plaques (OMT registry).
Minimal lumen area by Optical Coherence Tomography (OCT) | 4 years
  To establish the optimal OCT-derived minimal lumen area cutoff to predict an ischemic FFR in the non-culprit artery in the acute setting.
Accuracy of vulnerable plaque assessment by Optical Coherence Tomography (OCT) | 4 years
  To compare the agreement between local operators and the core-laboratory to assess vulnerable plaques by OCT.

CONTACTS AND LOCATIONS:
Locations (49):
- Spain (49):
  - Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitario A Coruña, A Coruña
  - Hospital General Universitario de Albacete, Albacete
  - Hospital General Universitario Dr.Balmis, Alicante
  - Hospital Universitari Sant Joan D'Alacant, Alicante
  - Hospital Universitari Germans Trias I Pujol, Badalona
  - Hospital Del Mar, Barcelona
  - Hospital de Santa Creu I Sant Pau, Barcelona
  - Hospital Universitari Vall Hebron, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Universitario Puerta Del Mar, Cadiz
  - Hospital General Universitario de Castellón, Castellon
  - Hospital General Universitario de Ciudad Real, Ciudad Real
  - Hospital Universitario Reina Sofia de Cordoba, Córdoba
  - Hospital General Universitario de Elche, Elche
  - Hospital Universitario de Cabueñes, Gijón
  - Hospital Universitario de Girona Dr Trueta, Girona
  - Hospital Universitario San Cecilio, Granada
  - Chu de Toledo, Guadalajara
  - Hospital Universitario Juan Ramon Jimenez, Huelva
  - H.U. de Gran Canaria-Dr. Negrin, Las Palmas de Gran Canaria
  - H.I.U. Materno Infantil de Las Palmas, Las Palmas de Gran Canaria
  - Hospital Universitario de Leon, León
  - Hospital La Princesa, Madrid
  - Hospital Universitario Gregorio Marañon, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Puerta de Hierro, Majadahonda
  - Hospital de Manises, Manises
  - Hospital de Merida, Mérida
  - Hospital Universitario Virgen Arrixaca, Murcia
  - Hospital Universitario Central de Asturias, Oviedo
  - Hospital Universitari Son Espases, Palma de Mallorca
  - Hospital Universitario de Navarra, Pamplona
  - Hospital Clinico Universitario de Salamanca, Salamanca
  - Hospital Universitario de Donostia, San Sebastián
  - Hospital Universitario Nuestra Señora de La Candelaria, Santa Cruz de Tenerife
  - Hospital Universitario Marqués de Valdecilla, Santander
  - Hospital Clinico Universitario de Santiago de Compostela, Santiago de Compostela
  - Hospital Universitario Virgen Del Rocio, Seville
  - Hospital Universitari Joan Xxiii, Tarragona
  - Hospital Universitari MútuaTerrassa, Terrassa
  - Hospital Universitario de Torrevieja, Torrevieja
  - Hospital Universitario 12 Octubre, Usera
  - Hospital Clinico Universitario de Valencia, Valencia
  - Hospital General Universitario de Valencia, Valencia
  - Hospital Universitari I Politecnic La Fe, Valencia
  - Hospital Clínico Universitario de Valladolid, Valladolid
  - Hospital Clinico Universitario Lozano Blesa, Zaragoza
  - Hospital Universitari Miquel Servet, Zaragoza

REFERENCES:
- [Background] Puymirat E, Cayla G, Simon T, Steg PG, Montalescot G, Durand-Zaleski I, le Bras A, Gallet R, Khalife K, Morelle JF, Motreff P, Lemesle G, Dillinger JG, Lhermusier T, Silvain J, Roule V, Labeque JN, Range G, Ducrocq G, Cottin Y, Blanchard D, Charles Nelson A, De Bruyne B, Chatellier G, Danchin N; FLOWER-MI Study Investigators. Multivessel PCI Guided by FFR or Angiography for Myocardial Infarction. N Engl J Med. 2021 Jul 22;385(4):297-308. doi: 10.1056/NEJMoa2104650. Epub 2021 May 16. PMID 33999545
- [Background] Mehta SR, Wood DA, Storey RF, Mehran R, Bainey KR, Nguyen H, Meeks B, Di Pasquale G, Lopez-Sendon J, Faxon DP, Mauri L, Rao SV, Feldman L, Steg PG, Avezum A, Sheth T, Pinilla-Echeverri N, Moreno R, Campo G, Wrigley B, Kedev S, Sutton A, Oliver R, Rodes-Cabau J, Stankovic G, Welsh R, Lavi S, Cantor WJ, Wang J, Nakamya J, Bangdiwala SI, Cairns JA; COMPLETE Trial Steering Committee and Investigators. Complete Revascularization with Multivessel PCI for Myocardial Infarction. N Engl J Med. 2019 Oct 10;381(15):1411-1421. doi: 10.1056/NEJMoa1907775. Epub 2019 Sep 1. PMID 31475795
- [Background] Erlinge D, Maehara A, Ben-Yehuda O, Botker HE, Maeng M, Kjoller-Hansen L, Engstrom T, Matsumura M, Crowley A, Dressler O, Mintz GS, Frobert O, Persson J, Wiseth R, Larsen AI, Okkels Jensen L, Nordrehaug JE, Bleie O, Omerovic E, Held C, James SK, Ali ZA, Muller JE, Stone GW; PROSPECT II Investigators. Identification of vulnerable plaques and patients by intracoronary near-infrared spectroscopy and ultrasound (PROSPECT II): a prospective natural history study. Lancet. 2021 Mar 13;397(10278):985-995. doi: 10.1016/S0140-6736(21)00249-X. PMID 33714389
- [Background] Stone GW, Maehara A, Ali ZA, Held C, Matsumura M, Kjoller-Hansen L, Botker HE, Maeng M, Engstrom T, Wiseth R, Persson J, Trovik T, Jensen U, James SK, Mintz GS, Dressler O, Crowley A, Ben-Yehuda O, Erlinge D; PROSPECT ABSORB Investigators. Percutaneous Coronary Intervention for Vulnerable Coronary Atherosclerotic Plaque. J Am Coll Cardiol. 2020 Nov 17;76(20):2289-2301. doi: 10.1016/j.jacc.2020.09.547. Epub 2020 Oct 15. PMID 33069847
- [Background] Denormandie P, Simon T, Cayla G, Steg PG, Montalescot G, Durand-Zaleski I, le Bras A, le Breton H, Valy Y, Schiele F, Cuisset T, Vanzetto G, Levesque S, Goube P, Nallet O, Angoulvant D, Roubille F, Charles Nelson A, Chatellier G, Danchin N, Puymirat E. Compared Outcomes of ST-Segment-Elevation Myocardial Infarction Patients With Multivessel Disease Treated With Primary Percutaneous Coronary Intervention and Preserved Fractional Flow Reserve of Nonculprit Lesions Treated Conservatively and of Those With Low Fractional Flow Reserve Managed Invasively: Insights From the FLOWER-MI Trial. Circ Cardiovasc Interv. 2021 Nov;14(11):e011314. doi: 10.1161/CIRCINTERVENTIONS.121.011314. Epub 2021 Aug 23. PMID 34420366
- [Derived] Gomez-Lara J, Lopez-Palop R, Rumiz E, Jurado-Roman A, Gomez-Menchero A, Valencia J, Fernandez E, Goncalves Ramirez LR, Brugaletta S, Millan R, Cortes C, Tejedor P, Gutierrez-Barrios A, Flores X, Cid-Alvarez AB, Garcia-Blas S, Garcia-Camarero T, Linares Vicente JA, Vaquerizo B, Cordoba Soriano JG, Caballero J, Cardenal Piris RM, Sanchez-Elvira G, Oyarzabal L, Pernigotti A, Tramullas A, Antuna P, Rodriguez-Leor O, Ojeda S, Rossello X, Gomez-Hospital JA, Bermejo J, Garcia-Garcia HM, Perez de Prado A, Gutierrez-Ibanes E. [Treatment of functionally nonsignificant vulnerable plaques in multivessel STEMI: design of the VULNERABLE trial]. REC Interv Cardiol. 2024 Jul 4;6(4):278-286. doi: 10.24875/RECIC.M24000468. eCollection 2024 Oct-Dec. PMID 40444169